CLINICAL TRIAL: NCT05035719
Title: Comparison Studies Comparing Hemodynamic Parameters Provided by the Caretaker
Brief Title: Comparison Studies Comparing Hemodynamic Parameters Provided by the Caretaker Against Respective Gold Standard References
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: CareTaker Medical LLC (Industry)
Collaborators: The Cooper Health System (Other)
Responsible Party: Sponsor
Other Study IDs: Hemo_002
Record Dates: First submitted 2021-08-31; First posted 2021-09-05 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Cardiac Output, Low
MeSH Terms: conditions — Cardiac Output, Low

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Group 1: Cardiac patients
  Interventions: Device: non-invasive cardiac output monitor

INTERVENTIONS:
Device: non-invasive cardiac output monitor — Equivalence of Caretaker cardiac output reading to reference standard
  Other Names: Equivalence of Caretaker cardiac output reading to reference standard

SUMMARY:
Comparison studies comparing hemodynamic parameters provided by the Caretaker against respective Gold Standard references.

DETAILED DESCRIPTION:
Comparison study comparing hemodynamic parameters provided by the Caretaker against respective Gold Standard references.

Specifically, continuous beat-by-beat blood pressure readings against arterial catheter readings and cardiac output (CO) and stroke volume (SV) measures against thermo-dilution measurements

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* able and willing to participate
* provide written consent

Exclusion Criteria:

* Unable to give written consent
* <18 years of age
* No or poor finger pulse, as determined through visual inspection for ischemic hands

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cardiac patients
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac output performance comparison | Change between several paired readings over the course of cardiac surgery (typically 2-4 hours)
  Comparison with thermo-dilution-based cardiac output, agreement within 1 l/min.

CONTACTS AND LOCATIONS:
Locations (1):
- Cooper University Hospital, Camden, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided